CLINICAL TRIAL: NCT04613492
Title: An Open-label, Phase 1 Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of MEDI9253, a Recombinant Newcastle Disease Virus Encoding Interleukin-12, in Combination With Durvalumab in Participants With Select Advanced/Metastatic Solid Tumors
Brief Title: A Study of MEDI9253 in Combination With Durvalumab in Select Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated early due to lack of efficacy and absence of biomarker evidence of MEDI9253's impact on the tumors.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D7880C00001; 2020-002294-96 (EudraCT Number)
Record Dates: First submitted 2020-10-28; First posted 2020-11-03 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Solid Tumors
Keywords: Solid Tumors
MeSH Terms: interventions — durvalumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- MEDI9253 Single Dose Level 1 + Durvalumab 1500 mg Q4W (Experimental): Participants will receive intravenous (IV) infusion of a single dose of MEDI9253 dose level 1 on Day 1. After 14 days (+7 days) of MEDI9253 dose, participants will receive IV durvalumab at 1500 mg once every 4 weeks (Q4W) until disease progression, clinical deterioration, withdrawal of consent, or unacceptable toxicity, for up to 2 years.
  Interventions: Biological: MEDI9253; Biological: Durvalumab
- MEDI9253 Single Dose Level 2 + Durvalumab 1500 mg Q4W (Experimental): Participants will receive IV infusion of a single dose of MEDI9253 dose level 2 on Day 1. After 14 days (+7 days) of MEDI9253 dose, participants will receive IV durvalumab at 1500 mg Q4W until disease progression, clinical deterioration, withdrawal of consent, or unacceptable toxicity, for up to 2 years.
  Interventions: Biological: MEDI9253; Biological: Durvalumab
- MEDI9253 Multiple Dose Level 2 + Durvalumab 1500 mg Q4W (Experimental): Participants will receive IV infusion of 3 weekly doses (±2 days) of MEDI9253 dose level 2 over a maximum of 17 days, with a minimum of 5 days between each dose. After 14 days (+7 days) post the last dose of MEDI9253, participants will receive IV durvalumab at 1500 mg Q4W until disease progression, clinical deterioration, withdrawal of consent, or unacceptable toxicity, for up to 2 years.
  Interventions: Biological: MEDI9253; Biological: Durvalumab
- MEDI9253 Multiple Dose Level 3 + Durvalumab 1500 mg Q4W (Experimental): Participants will receive IV infusion of 3 weekly doses (±2 days) of MEDI9253 dose level 3 over a maximum of 17 days, with a minimum of 5 days between each dose. After 14 days (+7 days) post the last dose of MEDI9253, participants will receive IV durvalumab at 1500 mg Q4W until disease progression, clinical deterioration, withdrawal of consent, or unacceptable toxicity, for up to 2 years.
  Interventions: Biological: MEDI9253; Biological: Durvalumab
- MEDI9253 Multiple Dose Level 3+Durva 1500 mg Q4W Seq 3A-DESENS (Experimental): Participants will receive IV infusion of 3 weekly doses (±2 days) of MEDI9253 dose level 3 over a maximum of 17 days, with a minimum of 5 days between each dose (first dose was administered at dose level 2 while second and third doses were administered at dose level 3). After 14 days (+7 days) post the last dose of MEDI9253, participants will receive IV durvalumab at 1500 mg Q4W until disease progression, clinical deterioration, withdrawal of consent, or unacceptable toxicity, for up to 2 years.
  Interventions: Biological: MEDI9253; Biological: Durvalumab
- MEDI9253 Multiple Dose Level 3+Durva 1500 mg Q4W Conc3B-DESENS (Experimental): Participants will receive IV infusion of 3 weekly doses (±2 days) of MEDI9253 dose level 3 over a maximum of 17 days, with a minimum of 5 days between each dose (first dose was administered at dose level 2 while second and third doses were administered at dose level 3) along with IV infusion of durvalumab 1500 mg Q4W starting from Day 8 (on the same day of second dose of MEDI9253) until disease progression, clinical deterioration, withdrawal of consent, or unacceptable toxicity, for up to 2 years.
  Interventions: Biological: MEDI9253; Biological: Durvalumab

INTERVENTIONS:
Biological: MEDI9253 — Participants will receive either single or multiple dose of MEDI9253; sequentially or concurrent with Durvalumab
Biological: Durvalumab — Participants will receive durvalumab treatment sequentially or concurrently with MEDI9253

SUMMARY:
Study D7880C00001 is a first-in-human (FIH), Phase 1, open-label, multicenter, dose escalation and dose expansion study to evaluate the safety, tolerability, PK, pharmacodynamics, and preliminary efficacy of MEDI9253 in combination with durvalumab in adult participants with select advanced/metastatic solid tumors.

DETAILED DESCRIPTION:
Up to approximately 192 participants may be assigned to study intervention in the study across approximately 30 sites globally.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be at least 18 years old at signing of informed consent.
2. Body weight > 35 kg at screening.

Exclusion Criteria:

1 Primary central nervous system (CNS) disease is excluded, as well as untreated or uncontrolled metastatic CNS involvement, leptomeningeal disease, or cord compression.

NOTE: CNS disease that has been treated and stable/controlled for at least 3 months is permitted. Participants with CNS disease controlled via systemic steroids are not permitted.

Ages: 18 Years to 101 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs) | Day 1 through 76.14 weeks (maximum observed duration)
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization, persistent or significant disability/incapacity, important medical event, congenital anomaly/birth defect (in the offspring of the subject). The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Number of Participants With Dose-limiting Toxicities (DLTs) | From the first dose of MEDI9253 through Day 14 (single dose cohorts) or Day 28 (multiple dose cohorts)
  DLT: Any study drug-related Grade (G) 3 or higher toxicity; aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥ 3 × upper limit of normal (ULN) together with total bilirubin (TBL) ≥ 2 × ULN; Grade ≥ 2 myocarditis; Grade 2 non-infectious pneumonitis that does not resolve to ≤ G 1 within 7 days; any ≥ G 2 MEDI9253-related toxicity that prevents the administration of more than 1 dose of MEDI9253; in the sequential dosing cohorts, any ≥ Grade 2 MEDI9253-related toxicity that prevents administration of the first dose of durvalumab; any AE that after consultation with the sponsor and investigators, is deemed to be a DLT.
Number of Participants With TEAEs Leading to Discontinuation | Day 1 through 76.14 weeks (maximum observed duration)
  Participants were permanently discontinued (PED) due to TEAE if: an AE that in the opinion of the investigator or the sponsor, warrants discontinuation of further dosing; an AE that met the criteria for a DLT during the DLT-evaluation period (from the first dose of MEDI9253 through Day 14 [single dose cohorts] or Day 28 [multiple dose cohorts]) unless criteria for initiation of durvalumab are met; an AE that required permanent discontinuation of study drug per toxicity management guidelines.
Number of Participants With Abnormal Vital Signs Reported as TEAEs | Day 1 through 76.14 weeks (maximum observed duration)
  Number of participants with abnormal vital signs reported as TEAEs are reported. Abnormal vital signs are defined as any abnormal finding in the vital sign parameters (body temperature, blood pressure, pulse oximetry [on MEDI9253 dosing days only], pulse rate, and respiratory rate).
Number of Participants With Abnormal Clinical Laboratory Parameters Reported as TEAEs | Day 1 through 76.14 weeks (maximum observed duration)
  Number of participants with abnormal clinical laboratory parameters reported as TEAEs are reported. Abnormal clinical laboratory parameters defined as any abnormal finding during analysis of hematology, clinical chemistry, coagulation, and urinalysis.
Number of Participants With Abnormal Electrocardiogram (ECG) Parameters Reported as TEAEs | Day 1 through 76.14 weeks (maximum observed duration)
  Number of participants with abnormal ECG reported as TEAEs are reported.
Number of Participants With Abnormal Physical Examination Reported as TEAEs | Day 1 through 76.14 weeks (maximum observed duration)
  Number of participants with abnormal physical examination reported as TEAEs are reported.

SECONDARY OUTCOMES:
Percentage of Participants With Objective Response (OR) According to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) | Baseline (Days -28 to -1) through 90 days post last dose (76.14 weeks)
  The OR is defined as confirmed complete response (CR) or confirmed partial response (PR) based on RECIST v1.1 criteria that occurs prior to the initiation of subsequent anticancer treatment and prior to progression. The CR is defined as disappearance of all target lesions (TLs) and non-target lesions (NTLs) present at baseline, any pathological lymph nodes selected as TLs or non-pathological lymph nodes of NTLs must have a reduction in short axis to < 10mm. The PR is defined as at least a 30% decrease in the sum of diameters of TLs, taking as reference the baseline sum of diameters as long as criteria for progressive disease (PD) are not met. PD is defined as "≥ 20% increase in the sum of diameters of TLs and an absolute increase of ≥ 5mm, taking as reference the smallest sum of diameters since treatment started including the baseline sum of diameters and unequivocal progression of existing NTLs. Percentage of participants with OR is reported.
Time to Response (TTR) According to RECIST V1.1 | Baseline (Days -28 to -1) through 90 days post last dose (76.14 weeks)
  The TTR is defined as the time from first dose until the first documentation of a subsequently confirmed OR. The OR is defined as confirmed CR or PR based on RECIST v1.1 criteria that occurs prior to the initiation of subsequent anticancer treatment and prior to progression. Only participants who have achieved confirmed CR or PR were evaluated for TTR. TTR was assessed using Kaplan-Meier methods.
Percentage of Participants With Disease Control Rate (DCR) at 16 Weeks According to RECIST v1.1 | Baseline (Days -28 to -1) through 90 days post last dose (76.14 weeks)
  The DCR at 16 weeks is defined as a best overall response of confirmed CR or PR or having stable disease (SD) (without subsequent cancer therapy) maintained for ≥ 15 weeks from first dose. SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD). PD is defined as a ≥ 20% increase in the sum of diameters of TLs and an absolute increase of ≥ 5mm, taking as reference the smallest sum of diameters since treatment started including the baseline sum of diameters. Percentage of participants who have disease control at 16 weeks is reported.
Progression Free Survival (PFS) According to RECIST v1.1 | Baseline (Days -28 to -1) through 90 days post last dose (76.14 weeks)
  The PFS is defined as the time from first dose until the date of first documented PD or death (by any cause in the absence of disease progression), regardless of whether the participant withdraws from study therapy or receives another anti-cancer therapy. Median number of months of PFS assessed via Kaplan-Meier method is reported. Here, number of participants analyzed denotes those participants who had PFS event.
Overall Survival (OS) | Baseline (Days -28 to -1) through 90 days post last dose (76.14 weeks)
  The OS is defined as the time from the date of first dose until death due to any cause regardless of whether the participant withdraws from study therapy or receives another anti-cancer therapy. Median number of months of OS assessed using Kaplan-Meier method is reported. Here, number of participants analyzed denotes those participants who had an event.
Whole Blood Viral Genome Concentrations of MEDI9253 for Single Dose Cohorts | Pre-dose, end of infusion (EOI); 1, 2, 4, 6, 9, 12, 24, 32, 40, 48, 72 hours and Days 7, 14, 21, 42 post EOI in Cycle 1 (each cycle is 28 days); and Durvalumab Cycle 3 pre-dose
  The whole blood viral genome concentrations of MEDI9253 for single dose cohorts are reported.
Whole Blood Viral Genome Concentrations of MEDI9253 for Multiple Dose Cohorts | Pre-dose, end of infusion, 1 day post dose on Days 1, 8, and 15; and 7 days post Dose 3; Durvalumab Cycle 1 (each cycle is 28 days)-Days 29, 36; Cycle 2-Days 36, 57; Cycle 3 Pre-dose Days 64, 85
  The whole blood viral genome concentrations of MEDI9253 for multiple dose cohorts are reported.
Plasma Interleukin (IL)-12 Concentrations for Single Dose Cohorts | Pre-dose, 1, 2, 4, 6, 9, 12, 24, 32, 40, 48, 72 hours and Days 7, 14, 21, 42 post end of infusion, and Durvalumab Cycle 3 (each cycle is 28 days) pre-dose
  The plasma IL-12 concentrations for single dose cohorts are reported.
Plasma IL-12 Concentrations for Multiple Dose Cohorts | Pre-dose, end of infusion, 1 day post dose on Days 1, 8, and 15; and 7 days post Dose 3; Durvalumab Cycle 1 (each cycle is 28 days)-Days 29, 36; Cycle 2-Days 36, 57; Cycle 3 Pre-dose Days 64, 85
  The plasma IL-12 concentrations for multiple dose cohorts are reported.
Cluster of differentiation (CD) 8 T cell Density as Assessed by Immunohistochemistry (IHC) | Baseline (Day -28 to -Day 1) and on Days 8, 15, 36, and 57
  The mean CD8 T cell density by IHC is reported.
Percentage of Programmed Cell Death Ligand 1 (PD-L1) Positive Tumor Cells by IHC | Baseline (Day -28 to -Day 1) and on Days 8, 15, 36, and 57
  The percentage of PD-L1 positive tumor cells by IHC is reported.
Percentage of Combined Tumor and Immune PD-L1 Positive Tumor Cells in Tumor Areas as Assessed by IHC | Baseline (Day -28 to -Day 1) and on Days 8, 15, 36, and 57
  The percentage of combined tumor and immune PD-L1 positive tumor cells in tumor areas as assessed by IHC is reported.
Number of Participants with Positive Neutralizing Antibody (nAb) Response to MEDI9253 | Baseline (pre-dose Day 1), Cycle 1 (each cycle is 28 days) Day 22, Cycle 2 Day 1, Cycle 3 Day 1, and 28 days after the last dose (7.47 weeks)
  Number of participants with positive nAb response to MEDI9253 is reported. Persistent positive is defined as positive at ≥ 2 post-baseline assessments (with ≥ 16 weeks between first and last positive) or positive at last post-baseline assessment. Transient positive is complement of persistent positive. Treatment boosted nAb is defined as baseline nAb titer that was boosted to a 4-fold or higher-level following study drug administration. Treatment emergent nAb is defined as the sum of treatment-induced nAb (post-baseline positive only) and treatment-boosted nAb.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (4):
  - Research Site, St Louis, Missouri
  - Research Site, Buffalo, New York
  - Research Site, New York, New York
  - Research Site, Pittsburgh, Pennsylvania
- France (3):
  - Research Site, Bordeaux
  - Research Site, Toulouse
  - Research Site, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7880C00001&attachmentIdentifier=bb5c95d0-de02-4682-9383-fc63571eaeb4&fileName=d7880c00001-study-synopsis-marked-for-redaction_Redacted.pdf&versionIdentifier=